CLINICAL TRIAL: NCT02549014
Title: A Single Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-1064
Brief Title: A Single Dose Study of the Safety, Pharmacokinetics and Pharmacodynamics of MK-1064 (MK-1064-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1064-001
Record Dates: First submitted 2015-09-11; First posted 2015-09-14 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Panel A: MK-1064 5 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 5 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel B: MK-1064 10 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 10 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel A: MK-1064 25 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 25 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel B: MK-1064 50 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 50 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel A: MK-1064 100 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 100 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel B: MK-1064 150 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 150 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel A: MK-1064 200 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 200 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel B: MK-1064 250 mg (Experimental): Within each of up to 4 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 250 mg in a fasted state. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: MK-1064
- Panel A: MK-1064 25 mg (Fed) (Experimental): In Period 5, participants received a single MK-1064 dose of 25 mg administered in the evening following a standard high-fat breakfast.
  Interventions: Drug: MK-1064
- Panel B: MK-1064 50 mg (Night) (Experimental): In Period 5, participants received a single MK-1064 dose of 50 mg administered in the evening after a 4-hour fast.
  Interventions: Drug: MK-1064
- Panels A & B: Placebo (Placebo Comparator): Within each of up to 5 treatment periods, 2 participants were randomly assigned to receive single oral doses of matching placebo in a fasted stated. There was to be a minimum 7-day washout between treatment periods for any given participant.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1064 — Dose for each period administered as oral MK-1064 tablets (1, 10 and 50 mg strengths)
  Arms: Panel A: MK-1064 100 mg; Panel A: MK-1064 200 mg; Panel A: MK-1064 25 mg; Panel A: MK-1064 25 mg (Fed); Panel A: MK-1064 5 mg; Panel B: MK-1064 10 mg; Panel B: MK-1064 150 mg; Panel B: MK-1064 250 mg; Panel B: MK-1064 50 mg; Panel B: MK-1064 50 mg (Night)
Drug: Placebo — Dose for each period administered as oral placebo tablets matching active MK-1064 tablets
  Arms: Panels A & B: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to evaluate the safety, pharmacokinetics and pharmacodynamics of rising, single oral doses MK-1064 in healthy, young, male participants. The primary pharmacokinetic hypothesis is that at least one dose of MK-1064 that is generally safe and well tolerated produces an average MK-1064 plasma concentration from 0 to 4 hours of ≥2.2 μM. Since this is an early Phase I assessment of MK-1064 in humans, the study protocol allows for modifications to the outlined dose, dosing regimen and/or clinical or laboratory procedures, if required to address study objectives and/or to ensure appropriate safety monitoring of participants.

DETAILED DESCRIPTION:
Two panels (Panels A and B), will receive alternating single rising oral doses of MK-1064/placebo (i.e., order of administration will be Panel A 5 mg, Panel B 10 mg, Panel A 25 mg, Panel B 50 mg, and continuing in this alternating sequence). Following dosing for a given treatment period, a minimum of 3 days will elapse before administration of the next scheduled dose. After administration of each dose, safety and tolerability will be reviewed. The decision to proceed to the next Panel/Period in the alternating sequence will be contingent on acceptable safety and tolerability data from the preceding Panels/Periods.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≤31 kg/m^2
* In good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests
* Nonsmoker and has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

* Mentally or legally incapacitated, significant emotional problems at screening or expected during the conduct of the study or history of a clinically significant psychiatric disorder within the last 10 years
* History of any persistent sleep abnormality (including difficulty falling asleep, difficulty staying asleep) lasting for 3 months or more, or history of obstructive sleep apnea, restless legs syndrome, or narcolepsy of any duration
* Participant has experienced poor quality sleep (including difficulty falling asleep, difficulty staying asleep) for at least 4 of 7 nights per week in the past 30 days prior to screening
* Participant works a night shift and is not able to avoid night shift work a minimum of 1 week before each treatment period
* Participant has traveled across 3 or more time zones (transmeridian travel) in the last 2 weeks prior to study
* Unwilling or unable to consume a standard high fat breakfast
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of seizures, epilepsy, stroke, peripheral neuropathy, or other clinically significant neurological disease or cognitive impairment
* History of cancer
* History of cataplexy
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies, beginning approximately 2 weeks prior to administration of the initial dose of study drug and throughout the study
* Participant consumes >3 servings of alcohol a day
* Participant consumes >6 caffeine servings a day
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to screening
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is currently a regular user of any illicit drugs or has a history of drug (including alcohol) abuse within 2 years of screening
* Is a regular user of sedative-hypnotic agents

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07-06 (Actual); Primary Completion 2009-09-29 (Actual); Study Completion 2009-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=1064-001&kw=1064-001&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male participants aged 18-45 years (inclusive) were recruited for this study.
Groups:
- Panel A: MK-1064: Panel A: Eight (8) participants were included in this panel. Within each of up to 5 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 and 2 participants were randomly assigned to receive single oral doses of matching placebo. MK-1064 was administered in rising single doses of 5, 25, 100 and 200 mg over Periods 1-4, in the morning with participants in a fasted condition. In Period 5, a single MK-1064 dose of 25 mg or placebo was administered to participants in the morning following a standard high-fat breakfast. Dosing periods alternated with Panel B. There was to be a minimum 7-day washout between treatment periods for any given participant.
- Panel B: MK-1064: Panel B: Eight (8) participants were included in this panel. Within each of up to 5 treatment periods, 6 participants were randomly assigned to receive single oral doses of MK-1064 and 2 participants were randomly assigned to receive single oral doses of matching placebo. MK-1064 was administered in rising single doses of 10, 50, 150 and 250 mg over Periods 1-4, in the morning with participants in fasted condition. In Period 5, a single MK-1064 dose of 50 mg or placebo was administered to participants in the evening after a 4-hour fast. Dosing periods alternated with Panel A. There was to be a minimum 7 day wash-out between treatment periods for any given participant.
Period: Overall Study
Arm/Group | Panel A: MK-1064 | Panel B: MK-1064
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-1064 | Panel B: MK-1064 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study drug, whether or not considered related to the use of study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of study drug, is also an AE.
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 60 days)
Population: All participants who received ≥1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- Panel A: MK-1064 25 mg (Fed): In Period 5, 6 participants received a single MK-1064 dose of 25 mg administered in the evening following a standard high-fat breakfast.
- Panel B: MK-1064 50 mg (Night): In Period 5, 6 participants received a single MK-1064 dose of 50 mg administered in the evening after a 4-hour fast.
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants | 4 | 5 | 5 | 5 | 5 | 5 | 6 | 6 | 3 | 3 | 5

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 1
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 60 days)
Population: All participants who received ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Average Plasma Concentration From Time Zero to 4 Hours (Area Under the Plasma Drug Concentration-time Curve From Time Zero to 4 Hours [AUC0-4hr]) Following Single Doses of MK-1064
Description: AUC0-4hr is the area under the plasma concentration-time curve from time 0 to 4 hours post-dose. This is a measure of the average amount of study drug (MK-1064) in the blood plasma over a period of 4 hours after the dose.
Time Frame: Pre-dose and 0.5, 1, 2, 3 and 4 hours post-dose
Population: All participants who received ≥1 dose of MK-1064.
Measure: Geometric Mean (Standard Deviation); unit: µmol*hr/L
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
µmol*hr/L | 0.77 (0.13) | 1.01 (0.42) | 2.99 (0.41) | 5.51 (2.29) | 9.75 (1.31) | 10.28 (3.42) | 20.12 (9.03) | 22.70 (7.98) | 1.61 (0.25) | 5.16 (2.60) |

4. Secondary Outcome: Area Under the Plasma Drug Concentration-time Curve From Time Zero to Last Measurable Concentration (AUC0-last) Following Single Doses of MK-1064
Description: AUC0-last is the area under the plasma concentration-time curve from time zero to time of last measurable concentration. It is is a measure of the amount of study drug (MK-1064) in the blood plasma from pre-dose until the last measurable concentration of study drug could be determined.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 48 hours post dose (all Periods); 72 hours post-dose (Periods 3 and 4 only)
Population: All participants who received ≥1 dose of MK-1064.
Measure: Geometric Mean (Standard Deviation); unit: µmol*hr/L
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
µmol*hr/L | 0.94 (0.25) | 1.67 (0.52) | 5.32 (0.71) | 9.89 (3.80) | 23.12 (6.23) | 25.92 (6.03) | 53.37 (13.78) | 57.10 (21.98) | 5.27 (1.13) | 9.91 (4.32) |

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single Doses of MK-1064
Description: Cmax is the maximum (peak) concentration of study drug (MK-1064) observed in blood plasma.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 48 hours post dose (all Periods); 72 hours post dose (Periods 3 and 4 only)
Population: All participants who received ≥1 dose of MK-1064.
Measure: Geometric Mean (Standard Deviation); unit: µmol/L
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
µmol/L | 0.37 (0.07) | 0.42 (0.16) | 1.06 (0.22) | 2.09 (0.77) | 3.60 (0.85) | 3.83 (1.46) | 6.78 (3.52) | 8.28 (2.87) | 0.80 (0.13) | 1.99 (0.64) |

6. Secondary Outcome: Time to Cmax (Tmax) Following Single Doses of MK-1064
Description: Tmax is the amount of time to reach maximum (peak) plasma drug concentration following drug administration.
Time Frame: as for outcome 5
Population: All participants who received ≥1 dose of MK-1064.
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
hr | 1.0 (0.07) [0.5 to 2.0] | 1.5 (0.16) [0.5 to 2.0] | 1.5 (0.22) [0.5 to 2.0] | 2.0 (0.77) [1.0 to 2.0] | 2.0 (0.85) [1.0 to 5.0] | 1.0 (1.46) [0.5 to 5.0] | 2.0 (3.52) [1.0 to 3.0] | 2.0 (2.87) [0.5 to 2.0] | 5.0 (0.13) [2.0 to 5.0] | 2.0 (0.64) [1.0 to 5.0] |

7. Secondary Outcome: Apparent Terminal Half-life (t1/2) Following Single Doses of MK-1064
Description: t1/2 is the elimination half-life of study drug. t1/2 is the time it takes for half of the study drug (MK-1064) in the blood plama to dissipate.
Time Frame: as for outcome 5
Population: All participants who received ≥1 dose of MK-1064.
Measure: Geometric Mean (Standard Deviation); unit: hr
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 0
hr | NA (NA) [0.5 to 2.0] — t1/2 estimates not available due to lack of data at terminal phase. | NA (NA) [0.5 to 2.0] — t1/2 estimates not available due to lack of data at terminal phase. | NA (NA) [0.5 to 2.0] — t1/2 estimates not available due to lack of data at terminal phase. | NA (NA) [1.0 to 2.0] — t1/2 estimates not available due to lack of data at terminal phase. | 11.1 (5.0) [1.0 to 5.0] | 6.8 (3.2) [0.5 to 5.0] | 7.5 (1.6) [1.0 to 3.0] | 8.6 (2.7) [0.5 to 2.0] | NA (NA) [2.0 to 5.0] — t1/2 estimates not available due to lack of data at terminal phase. | NA (NA) [1.0 to 5.0] — t1/2 estimates not available due to lack of data at terminal phase. |

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 60 days)
Description: All participants who recieved ≥1 dose of study drug. Adverse events are reported based on the study drug a participant was taking at the time of the event.
Arm/Group | Panel A: MK-1064 5 mg | Panel B: MK-1064 10 mg | Panel A: MK-1064 25 mg | Panel B: MK-1064 50 mg | Panel A: MK-1064 100 mg | Panel B: MK-1064 150 mg | Panel A: MK-1064 200 mg | Panel B: MK-1064 250 mg | Panel A: MK-1064 25 mg (Fed) | Panel B: MK-1064 50 mg (Night) | Panels A & B: Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 5/6 | 5/6 | 5/6 | 5/6 | 6/6 | 6/6 | 3/6 | 3/6 | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-1064 5 mg (N=6) | Panel B: MK-1064 10 mg (N=6) | Panel A: MK-1064 25 mg (N=6) | Panel B: MK-1064 50 mg (N=6) | Panel A: MK-1064 100 mg (N=6) | Panel B: MK-1064 150 mg (N=6) | Panel A: MK-1064 200 mg (N=6) | Panel B: MK-1064 250 mg (N=6) | Panel A: MK-1064 25 mg (Fed) (N=6) | Panel B: MK-1064 50 mg (Night) (N=6) | Panels A & B: Placebo (N=16)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-1064 5 mg (N=6) | Panel B: MK-1064 10 mg (N=6) | Panel A: MK-1064 25 mg (N=6) | Panel B: MK-1064 50 mg (N=6) | Panel A: MK-1064 100 mg (N=6) | Panel B: MK-1064 150 mg (N=6) | Panel A: MK-1064 200 mg (N=6) | Panel B: MK-1064 250 mg (N=6) | Panel A: MK-1064 25 mg (Fed) (N=6) | Panel B: MK-1064 50 mg (Night) (N=6) | Panels A & B: Placebo (N=16)
Sensation of block in ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloated feeling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tiredness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fractured thumb (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scalp laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thumb sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Painful L arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowsiness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental concentration difficulty (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 5 (5) | 5 (5) | 6 (6) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.